# Statistical Analysis Plan B5K-EW-IBHG

Comparative Pharmacokinetics and Pharmacodynamics of Human Regular U-500 Insulin Administered Subcutaneously as a Bolus via Syringe versus Continuous Subcutaneous Insulin Infusion and Characterization of TID and BID Dosing at Steady State in High-Dose Insulin-Treated Subjects with Type 2 Diabetes Mellitus

NCT02588950

Approval Date: 21-Sep-2015

# STATISTICAL ANALYSIS PLAN

Comparative Pharmacokinetics and Pharmacodynamics of Human Regular U-500 Insulin Administered Subcutaneously as a Bolus via Syringe versus Continuous Subcutaneous Insulin Infusion and Characterization of TID and BID Dosing at Steady State in High-Dose Insulin-Treated, Obese Subjects with Type 2 Diabetes Mellitus

Statistical Analysis Plan Status: Final Statistical Analysis Plan Date: 15-September-2015

Study Drug: LY041001

Sponsor Reference: B5K-EW-IBHG Covance CRU Study: 1000071-8316164

Clinical Phase I

Approval Date: 21-Sep-2015 GMT

# 1. TABLE OF CONTENTS

| 1. | TABLE OF CONTENTS | 2 |
|-----------|------------------------------------------------------------|----|
| 2. | ABBREVIATIONS | 3 |
| 3. | INTRODUCTION | 5 |
| 4. | STUDY OBJECTIVES | 5 |
| | Primary Objectives | 5 |
| | Secondary Objectives | 6 |
| | Exploratory Objectives | 6 |
| 5. | STUDY DESIGN | 6 |
| 6. | TREATMENTS | 7 |
| <b>7.</b> | SAMPLE SIZE JUSTIFICATION | 7 |
| 8. | DEFINITION OF ANALYSIS POPULATIONS | 8 |
| 9. | STATISTICAL METHODOLOGY | 8 |
| | 9.1 General. | 8 |
| | 9.2 Demographics and Subject Disposition | 8 |
| | 9.3 Pharmacokinetic Assessment | 9 |
| | 9.3.1 Pharmacokinetic Analysis | 9 |
| | 9.3.2 Pharmacokinetic Statistical Methodology | 10 |
| | 9.4 Pharmacodynamic Assessment | 10 |
| | 9.4.1 Pharmacodynamic Analysis | 10 |
| | 9.4.2 Pharmacodynamic Statistical Methodology | 11 |
| | 9.5 Safety and Tolerability Assessments | 11 |
| | 9.5.1 Adverse events | 11 |
| | 9.5.2 Concomitant medication | 12 |
| | 9.5.3 Clinical laboratory parameters | 12 |
| | 9.5.4 Vital signs | 12 |
| | 9.5.5 Blood Glucose Monitoring and Hypoglycemia | 12 |
| | 9.5.6 Other assessments. | 12 |
| | 9.5.7 Safety and Tolerability Statistical Methodology | 12 |
| 10 | ). INTERIM ANALYSES | 13 |
| 11 | . CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES | 13 |
| | 2. REFERENCES | |
| 13 | 3. DATA PRESENTATION | 13 |
| | 13.1 Derived Parameters | 13 |
| | 13.2 Missing Data | 13 |
| | 13.3 Insufficient Data for Presentation | 13 |

### 2. ABBREVIATIONS

Abbreviations pertain to the Statistical Analysis Plan (SAP) only (not the tables, figures and listings [TFLs]).

AE Adverse event

AUC Area under the concentration versus time curve

AUC(0-t<sub>last</sub>) Area under the concentration versus time curve from time zero to

time t, where t is the last time point with a measurable concentration

BID Twice daily

BQL Below the quantifiable lower limit of the assay

C<sub>max</sub> Maximum observed drug concentration

CI Confidence interval

CL/F Apparent total body clearance of drug calculated after extra-vascular

administration

CRF Case Report Form

CSR Clinical Study Report

CSII Continuous subcutaneous insulin infusion

CRU Clinical Research Unit
CV Coefficient of variation

Early  $tR_{max50}$  Time of 50% of maximum GIR before  $R_{max}$ 

ECB Early clinical biometrics

ECG Electrocardiogram

e.g. For example (Latin: *exempli gratia*)

GIR Glucose infusion rate

ICH International Conference on Harmonisation Late  $tR_{max50}$  Time of 50% of maximum GIR after  $R_{max}$ 

LLOQ Lower limit of quantitation

LS Least square

MDI Multiple daily injections

MedDRA Medical Dictionary for Regulatory Activities

NA Not applicable

PD Pharmacodynamic

PK Pharmacokinetic

QTcB QT interval corrected using Bazett's formula

QTcF QT interval corrected using Fridericia's formula

R<sub>max</sub> Maximum glucose infusion rate

SAP Statistical Analysis Plan

SC Subcutaneous

SD Standard deviation

SMPG Self-monitored plasma glucose

TDD Total daily dose

T2DM Type 2 diabetes mellitus

TID Thrice daily

TFLs Tables, Figures, and Listings

 $t_{1/2}$  Half-life associated with the terminal rate constant ( $\lambda_z$ ) in non-

compartmental analysis

t<sub>max</sub> Time of maximum observed drug concentration

tR<sub>max</sub> Time of maximum glucose infusion rate

 $V_z/F$  Apparent volume of distribution during the terminal phase after

extra-vascular administration

WHO World Health Organization

## 3. INTRODUCTION

This SAP has been developed after review of the Clinical Study Protocol (final version dated 29 April 2015 and amendment (a) dated 24 August 2015).

This SAP describes the planned analysis of the safety, tolerability and pharmacokinetic (PK) and pharmacodynamic (PD) data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical and PK analyses of data. In general, the analyses are based on information from the protocol, unless they have been modified by agreement between Eli Lilly and Company and Covance Early Clinical Biometrics (ECB). A limited amount of information concerning this study (e.g., objectives, study design) is given to help the reader's interpretation. This SAP must be signed off prior to first subject administration for this study. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified in the CSR. Any substantial deviations from this SAP will be agreed upon between Eli Lilly and Company and Covance ECB and identified in the CSR. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

### 4. STUDY OBJECTIVES

## **Primary Objectives**

Part A: to compare the  $t_{max}$  of a 100-U bolus of U-500R (500 U/mL) administered via single subcutaneous (SC) injection versus a 100-U bolus of U-500R administered via continuous subcutaneous insulin infusion (CSII) in high-dose insulin-treated, obese subjects with type 2 diabetes mellitus (T2DM).

Part B: to evaluate the area under the concentration versus time curve (AUC) from time zero to 24 hours postdose (AUC[0-24]), maximum drug concentration ( $C_{max}$ ), and maximum glucose infusion rate ( $R_{max}$ ) of U-500R at steady state following thrice daily (TID) or twice daily (BID) SC dosing in the study population.

## **Secondary Objectives**

Part A: to compare the time of maximum glucose infusion rate (GIR) (tR<sub>max</sub>) and exposure (AUC from time zero to time t, where t is the last time point with a measurable concentration [AUC(0-t<sub>last</sub>)]) of a 100-U bolus of U-500R administered via single SC injection versus CSII in the study population.

Part B: to evaluate the time of  $C_{max}$  ( $t_{max}$ ), total amount of glucose infused ( $G_{tot}$ ) and  $tR_{max}$  of U-500R at steady state following TID or BID SC dosing in the study population.

## **Exploratory Objectives**

Other PK and PD parameters may be evaluated including but not limited to:

Part A: half-life associated with the terminal rate constant in no ncompartmental analysis ( $t_{1/2}$ ), apparent total body clearance of drug calculated after extra -vascular administration (CL/F), and apparent volume of distribution during the terminal phase after extra -vascular administration ( $V_z$ /F), time of last GIR measurement ( $tR_{last}$ ), the time of first change of GIR postdose ( $tR_{onset}$ ), the time of 50% of maximum GIR before  $R_{max}$  (early  $tR_{max50}$ ), and the time of 50% of maximum GIR after  $R_{max}$  (late  $tR_{max50}$ ) in the study population.

Part B: AUC of U-500R over each dosing interval and over each meal at steady state following TID or BID SC dosing in the study population.

### 5. STUDY DESIGN

This is a 2-part, Phase 1 (postmarketing), single-center, 3-period, 4-sequence, randomized, open-label, crossover euglycemic clamp study in high-dose insulin-treated, obese subjects with T2DM. Part A (Periods 1 and 2) will compare the PK and PD of a 100-U bolus of U-500R administered via single SC injection versus a 100-U bolus of U-500R administered via CSII. Subjects completing Part A will transition to Part B (Period 3), which will evaluate the PK and PD characteristics of U-500R administered by TID and BID multiple daily injections (MDIs) under steady-state conditions.

Up to 32 subjects may be enrolled to achieve a target of approximately 24 completing all 3 periods of the study.

Subjects will be randomly assigned to 1 of 4 dosing sequences (Table 1.). Each subject will be administered 100 U of U-500R by single SC injection, and 100 U of U-500R by CSII in Part A and either TID U-500R or BID U-500R in Part B.

| Table | 1. | D | osing | Sc | hec | lule | • |
|--------|----|--------------------|--------|---------------|-------|------|---|
| 1 abic | 1. | $\boldsymbol{\nu}$ | USILIE | $\mathcal{S}$ | .1166 | ıuı | _ |

| | Part A | | Part B |
|----------|----------|----------|----------|
| Sequence | Period 1 | Period 2 | Period 3 |
| 1 | SC | CSII | TID |
| 2 | CSII | SC | BID |
| 3 | SC | CSII | BID |
| 4 | CSII | SC | TID |

Abbreviations: BID=twice-daily administration of U-500R; CSII=100 U U-500R administered via continuous subcutaneous insulin infusion; SC=100 U U-500R administered via single subcutaneous injection; TID=thrice-daily administration of U-500R



Figure 1. Study Design

#### 6. TREATMENTS

The following is a list of the study treatment abbreviations that will be used in the TFLs.

| Study Treatment Name | Treatment order in TFL |
|---------------------------|------------------------|
| 100-U bolus U-500R (SC) | 1 |
| 100-U bolus U-500R (CSII) | 2 |
| U-500R (BID) | 3 |
| U-500R (TID) | 4 |

## 7. SAMPLE SIZE JUSTIFICATION

The primary objective of Part A of the study is to compare the t max of U-500R administered by single SC injection or CSII. Up to 32 subjects may be enrolled to ensure that approximately 24 subjects complete the study.

The sample size is based on a calculation of precision of the  $t_{max}$ . Intra-subject variability for  $t_{max}$  has not been assessed previously. Based on an assumption of an intra-subject variability estimate of 20% for  $t_{max}$ , a sample size of 24 completed subjects in Part A will provide approximately 90% coverage probability that the half-width of the 90% confidence interval (CI) for the ratio of

geometric means for  $t_{\text{max}}$  will be within 0.116 in the log scale, which corresponds to approximately 12% of the geometric mean ratio estimate in the natural scale.

If any subjects discontinue the study prior to completion of the 3 periods, the replacement subjects who are enrolled will assume the discontinued subjects' randomization schedule and will complete all 3 periods.

### 8. DEFINITION OF ANALYSIS POPULATIONS

The "Safety" population will consist of all subjects who received at least one dose of study drug, and have at least one postdose safety assessment.

The "Pharmacokinetic" population will consist of all subjects who received at least one dose of study drug and have evaluable PK data.

The "Pharmacodynamic" population will consist of all subjects who received at least one dose of study drug and have evaluable PD data.

All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when subjects are assigned to analysis populations.

## 9. STATISTICAL METHODOLOGY

### 9.1 General

Data listings will be provided for all data that is databased. Summary statistics and statistical analysis will only be presented for data where detailed in this SAP. For continuous data, summary statistics will include the arithmetic mean, arithmetic standard deviation (SD), median, min, max and N; for log-normal data (e.g. the PK parameters: AUCs and C<sub>max</sub>) the geometric mean and geometric coefficient of variation (CV%) will also be presented. For categorical data, frequency count and percentages will be presented. Data listings will be provided for all subjects up to the point of withdrawal, with any subjects excluded from the relevant population highlighted. Summary statistics and statistical analyses will generally only be performed for subjects included in the relevant analysis population.

Mean change from baseline is the mean of all individual subjects' change from baseline values. Each individual change from baseline will be calculated by subtracting the individual subject's baseline value from the value at the timepoint. The individual subject's change from baseline values will be used to calculate the mean change from baseline using a SAS procedure such as Proc Univariate.

The TFLs will be programmed using SAS® Version 9.3 or greater.

## 9.2 Demographics and Subject Disposition

Subject disposition will be listed. The demographic variables age, sex, race, ethnicity, country of enrollment, site ID, body weight, height and body mass index will be summarized and listed.

Screening HbA1c, HbA1c > 8.0%, HbA1c  $\leq 8.0\%$ , fasting blood glucose, duration of T2DM and prestudy insulin treatment will be summarized and listed.

### 9.3 Pharmacokinetic Assessment

## 9.3.1 Pharmacokinetic Analysis

For the primary analysis, serum immunoreactive concentrations of insulin will be corrected using C-peptide data. Specifically, drug insulin concentrations will be calculated as the difference between total insulin and endogenous insulin, which in turn will be estimated with the C-peptide concentration data using Owens method (Owens 1986) with the following equation:

Drug insulin = Total insulin – 
$$F*C$$
-peptide

where F is the average of the ratios of insulin to C-peptide at baselines (-0.5, and 0 hour) and will be calculated for the subject per the following rule:

- 1. If there is BQL values for insulin or C-peptide, set them to ½ LLOQ.
- 2. Take the mean of the ratios of insulin to C-peptide at the two pre-dose time points (-0.5h, and 0h) during the single SC injection period as the F for the subject.

Pharmacokinetic parameter estimates will be calculated using non-compartmental methods of analysis in validated software (Phoenix WinNonlin Version 6.3, Pharsight Corporation, USA or later). The analyses will be performed according to the Lilly Global Pharmacokinetics, Pharmacodynamics, and Pharmacometrics Divisional Standard Operating Procedures. The actual validated software version used when actual analyses are conducted will be specified in the clinical study report. C-peptide may be used to correct serum immunoreactive insulin concentrations for endogenous insulin.

The primary parameter for analysis in Part A will be  $t_{max}$ . Other noncompartmental parameters such as  $C_{max}$ , AUC from time zero to infinity (AUC[0- $\infty$ ]), AUC(0- $t_{last}$ ), half-life associated with the terminal rate constant in noncompartmental analysis ( $t_{1/2}$ ), the last time point with a measurable concentration ( $t_{last}$ ), apparent total body clearance of drug calculated after extravascular administration (CL/F), and apparent volume of distribution during the terminal phase after extra-vascular administration ( $V_z/F$ ) may be reported, as appropriate.

In the treatment of CSII, the PK profile of insulin via SC injection can be corrected by subtracting baseline concentration, given steady-state of infused basal insulin via CSII will be reached after 12hrs.

The primary PK parameters for Part B will be AUC(0-24) and  $C_{max}$ ; other PK parameters such as  $t_{max}$  and AUC of U-500R over each dosing interval and over each assumed meal time period at steady state may also be reported, as appropriate.

Parameters will be individually calculated by Eli Lilly and Company and sent to Covance for statistical analysis.

## 9.3.2 Pharmacokinetic Statistical Methodology

For Part A, the primary parameter for statistical analysis will be  $t_{max}$ . The values for  $t_{max}$  will be log-transformed and evaluated in a linear mixed-effects model with fixed effects for administration method, period and sequence order (order 1 is derived based on sequences 1 and 3, and order 2 is derived based on sequences 2 and 4), and a random effect for subject. The difference in least squares (LS) means along with the 90% CI will be back-transformed to present the ratios of geometric means and the 90% CI for the comparison of the administration methods (single SC injection [test] and CSII [reference]). This same analysis will be repeated for  $AUC(0-t_{last})$ ,  $AUC(0-\infty)$ , and  $C_{max}$ .

## Example SAS code:

```
proc mixed data= ;
  class seqorder period method subject;
  model l_pk = seqorder period method / outpred=resids ddfm=kr;
  random subject;
  lsmeans method / pdiff alpha=0.1;
  ods output lsmeans=lsm;
  ods output diffs=diff;
run; quit;
```

The values of  $t_{max}$  will also be analyzed non-parametrically using a Wilcoxon signed-rank test using the SAS procedure PROC UNIVARIATE. Median differences and approximate 90% CIs for the difference will be calculated for the comparisons of the administration methods (single SC injection and CSII).

No formal statistical analysis will be conducted for Part B.

PK parameters will be listed and summarized for both parts of the study.

## 9.4 Pharmacodynamic Assessment

### 9.4.1 Pharmacodynamic Analysis

The PD measurements will be derived from the euglycemic clamp procedure, where the glucose infusion rate (GIR) over time is used as a measure of insulin effect. The analyses will be performed according to the Lilly Global PK, PD, and Pharmacometrics Divisional Standard Operating Procedures.

A locally weighted scatterplot smoothing (LOESS) function will be applied to all individual GIR versus time profiles in each treatment group using S Plus® software (Version 8.2 or higher, TIBCO, USA). The fitted data for each subject will be used to calculate the PD parameters: the maximum GIR ( $R_{max}$ ), the total amount of glucose infused ( $G_{tot}$ ) over the duration of the clamp procedure, the time of maximum GIR ( $tR_{max}$ ). Raw (that is, observed) GIR values from each clamp procedure will be used to calculate other PD parameters, such as the time of first change of GIR postdose ( $tR_{onset}$ ), the time of last measurable GIR ( $tR_{last}$ ). Other parameters, such as early  $tR_{max50}$ , and late  $tR_{max50}$ , may also be reported. Parameters will be individually calculated by Eli Lilly and Company and sent to Covance for statistical analysis.

## 9.4.2 Pharmacodynamic Statistical Methodology

For Part A, the values of tR<sub>max</sub> will be analyzed non-parametrically using a Wilcoxon signed-rank test using the SAS procedure PROC UNIVARIATE. Median differences and approximate 90% CIs for the difference will be calculated for the comparisons of the administration methods (single SC injection [test] and CSII [reference]).

The PD parameters ( $R_{max}$  and  $G_{tot}$ ) will be log-transformed prior to analysis and a linear mixed-effects model fitted to the data, with administration method, period, and sequence order (order 1 is derived based on sequences 1 and 3, and order 2 is derived based on sequences 2 and 4), as fixed effects and subject as a random effect. For each parameter, the difference in LS means along with the 90% CI will be back-transformed to present the ratios of geometric means and the CI for comparison of the administration methods.

See the PK statistical methodology for example SAS code.

Other time parameters ( $tR_{last}$ ,  $tR_{onset}$ , early  $tR_{max50}$ , and late  $tR_{max50}$ ) will be analyzed non-parametrically if reported.

No formal statistical analysis will be conducted for Part B.

PD parameters will be listed and summarized for both parts of the study.

Mean daily 4-point self-monitored plasma glucose (SMPG) data will be listed and also summarised for the 5 days prior to period 1, 2 and 3. Figures of mean SMPG prior to periods 1, 2 and 3 will be produced. Profiles prior to meals, bedtime and at 3am will also be produced as appropriate.

Exploratory analyses may be performed for other PD parameters as deemed appropriate.

## 9.5 Safety and Tolerability Assessments

#### 9.5.1 Adverse events

Where changes in severity are recorded in the Case Report Form (CRF), each separate severity of the adverse event (AE) will be reported in the listings, only the most severe will be used in the summary tables. A pre-existing condition is defined as an AE that starts before the subject has provided written informed consent and is ongoing at consent. A non-treatment emergent AE is defined as an AE which starts after informed consent but prior to dosing. A treatment-emergent AE is defined as an AE which occurs postdose or which is present prior to dosing and becomes more severe postdose.

All AEs will be listed. Treatment-emergent AEs will be summarized by treatment, severity and relationship to the study drug. The frequency (the number of adverse events, the number of subjects experiencing an adverse event and the percentage of subjects experiencing an adverse event) of treatment-emergent adverse events will be summarized by treatment, Medical Dictionary for Regulatory Activities (MedDRA) version 18.0 system organ class and preferred

term. The summary and frequency adverse event tables will be presented for all causalities and those considered related to the study drug. Any serious adverse events will be tabulated.

### 9.5.2 Concomitant medication

Concomitant medication will be coded using the WHO drug dictionary (Version March 2015). Concomitant medication and anti-hyperglycemic concomitant medication will be listed.

## 9.5.3 Clinical laboratory parameters

All clinical chemistry, hematology and urinalysis data will be listed. Additionally, clinical chemistry, hematology and urinalysis data outside the reference ranges will be listed.

Values for any clinical chemistry, hematology and urinalysis values outside the reference ranges will be flagged on the individual subject data listings.

## 9.5.4 Vital signs

Vital signs data will be summarized by treatment together with changes from baseline, where baseline is defined as Day 1 predose of the relevant period. Figures of mean vital signs and change from baseline profiles will be presented. Furthermore, values for individual subjects will be listed.

## 9.5.5 Blood Glucose Monitoring and Hypoglycemia

Hypoglycemic events will be appropriately recorded in the CRF.

In the case of a hypoglycemic event, the actual blood glucose value, if measured, will be recorded in the CRF, together with any treatments administered.

Hypoglycemic events will be listed, and summarised if appropriate. Severe hypoglycemic events will be reported as SAEs.

#### 9.5.6 Other assessments

Body weight will be listed. Change in weight and BMI from period 1 to period 2, and from period 2 to period 3 will be listed and summarized.

Change in total daily dose (Units and Units/kg) from pre-Period 3 U-100 to Period 3 U-500R will be listed.

All other safety assessments not detailed in this section will be listed but not summarized or statistically analyzed.

### 9.5.7 Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

## 10. INTERIM ANALYSES

An interim analysis will be conducted after approximately 12 subjects have completed both periods of Part A of the study. An interim analysis of safety, PK and PD will be carried out and will be used to inform ongoing analysis of a Phase 3b trial, as appropriate.

### 11. CHANGES FROM THE PROTOCOL SPECIFIED STATISTICAL ANALYSES

There were no changes from the protocol specified statistical analyses.

### 12. REFERENCES

- 1. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Statistical Principles for Clinical Trials (E9), 5 February 1998.
- 2. International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use, ICH Harmonized Tripartite Guideline, Structure and Content of Clinical Study Reports (E3), 30 November 1995.
- 3. DR Owens, ed. Human Insulin: Clinical pharmacological studies in normal man. Lancaster, UK: MTP Press; 1986.

#### 13. DATA PRESENTATION

#### 13.1 Derived Parameters

Individual derived parameters (e.g. PK parameters) and appropriate summary statistics will be reported to three significant figures. Observed concentration data, e.g.  $C_{max}$ , should be reported as received. Observed time data, e.g.  $t_{max}$ , should be reported as received. N and percentage values should be reported as whole numbers. Median values should be treated as an observed parameter and reported to the same number of decimal places as minimum and maximum values.

## 13.2 Missing Data

Missing data will not be displayed in listings.

### 13.3 Insufficient Data for Presentation

Some of the TFLs may not have sufficient numbers of subjects or data for presentation. If this occurs, the blank TFL shell will be presented with a message printed in the centre of the table, such as, "No serious adverse events occurred for this study."

Leo Document ID = e2cae2d2-b284-432e-b2c9-747f48e1b68b

Approver: PPD

Approval Date & Time: 18-Sep-2015 08:44:08 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 18-Sep-2015 14:07:07 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 21-Sep-2015 08:47:33 GMT

Signature meaning: Approved